CLINICAL TRIAL: NCT02272517
Title: An Interventional, Randomised, Double-blind, Parallel-group, Active-comparator, Flexible-dose Study on the Efficacy of Vortioxetine Versus Escitalopram on Cognitive Dysfunction in Patients With Inadequate Response to Current Antidepressant Treatment of Major Depressive Disorder
Brief Title: Efficacy of Vortioxetine Versus Escitalopram on Cognitive Function in Patients With Inadequate Response to Current Antidepressant Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15907A; 2014-000231-16 (EudraCT Number)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
Keywords: Vortioxetine; Cognition
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram 10-20 mg (Active Comparator): Encapsulated tablets once daily for 8 weeks
  Interventions: Drug: Escitalopram 10-20 mg
- Vortioxetine 10-20 mg (Experimental): Encapsulated tablets once daily for 8 weeks
  Interventions: Drug: Vortioxetine 10-20 mg

INTERVENTIONS:
Drug: Vortioxetine 10-20 mg
  Other Names: Brintellix®; Lu AA21004
  Arms: Vortioxetine 10-20 mg
Drug: Escitalopram 10-20 mg
  Arms: Escitalopram 10-20 mg

SUMMARY:
This study aims at evaluating the effect of vortioxetine on cognitive dysfunction in major depressive disorder (MDD) patients with inadequate response to current antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has MDD, diagnosed according to DSM-IV-TR™ recurrent MDE (classification 296.3x) as confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has depressive symptoms currently considered as non- or only partially responsive (inadequate response), to one adequate course of SSRI/SNRI antidepressant monotherapy and is candidate for a switch in the investigator's opinion.
* The patient wants to stop taking his/her current SSRI/SNRI treatment due to inadequate response confirmed by the Antidepressant Treatment Response Questionnaire (ATRQ), <50% response to current treatment).
* The patient must have been treated by SSRI/SNRI monotherapy (citalopram, paroxetine, sertraline, duloxetine, or venlafaxine) for at least 6 weeks at licensed doses prior to the Screening Visit.
* The patient has a PHQ-9 total score ≥14.
* The patient has a MADRS total score ≥ 22.
* The patient has had the current MDE for ≤1 year.
* The patient has a Perceived Deficits Questionnaire - Depression (PDQ-D) total score >25.
* The patient is a man or woman aged ≥18 and ≤65 years.

Exclusion Criteria:

* The patient has a score ≥70 on the DSST (Number of Correct Symbols) at the Baseline Visit.
* The patient has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* The patient has any current psychiatric disorder or Axis I disorder (according to DSMIV-TR™ criteria) other than MDD, as assessed using MINI.
* The patient has a current or has had a diagnosis of dysthymic disorder within 3 months preceding the onset of current episode (DSM-IV-TR™ criteria).
* The patient has borderline, schizotypal, schizoid, paranoid, histrionic, antisocial personality disorders (axis II) as comorbid or primary diagnosis (DSM-IV-TR™ criteria).
* The patient has history of previous MDEs considered as treatment resistant defined as inadequate response (incomplete or no therapeutic response) to two prior courses of at least 6 weeks of conventional antidepressant drugs in adequate dosages or, the patient has treatment-resistant depression in the investigator's judgement.
* The patient suffers from personality disorders, mental retardation, pervasive development disorder, attention-deficit/hyperactivity disorder, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient has a diagnosis of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) (DSM-IV-TR™ criteria) that has not been in sustained full remission at least 2 years prior to the Screening Visit.
* The patient has a current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features (DSM-IV-TR™ criteria).

Other protocol defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Digit Symbol Substitution Test (DSST) | Baseline to Week 8
  The DSST is recognised as covering all of the cognitive performance aspects: speed of processing, executive functioning, and attention

SECONDARY OUTCOMES:
Change in Rey Auditory Verbal Learning Test (RAVLT) | Baseline to Week 8
  Learning [acquisition] and memory [delayed recall])
Change in Trail Making Test A (TMT-A) | Baseline to Week 8
  Speed of processing
Change in Trail Making Test B (TMT-B) | Baseline to Week 8
  Executive functioning
Change in Reaction time score; CRT attention | Baseline to Week 8
Change in reaction time score SRT - simple reaction time | Baseline to week 8
Change in STROOP incongruent score | Baseline to Week 8
  Executive functioning
Change in STROOP congruent score | Baseline to Week 8
  Speed of processing
Change in Perceived Deficits Questionnaire - Depression (PDQ-D) total score | Baseline to Week 8
  Patient-reported cognitive function outcome including attention concentration, retrospective memory, prospective memory, and, planning organization
Change in Patient Health Questionnaire-9 (depressive symptoms) (PHQ-9) total score | Baseline to Week 8
  Patient-reported outcome
Change in Clinical Global Improvement - Severity (CGI-S) | Baseline to Week 8
Clinical Global Improvement (CGI-I) | Week 8
Change in Functioning Assessment Short Test (FAST) | Baseline to Week 8
Change in University of San Diego Performance-based Skills Assessment - Brief (UPSA-B) total score | Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (16):
- Finland (5):
  - FI005, Helsinki
  - FI001, Kuopio
  - FI006, Kupio
  - FI007, Tampere
  - FI004, Turku
- Germany (2):
  - DE005, Bochum
  - DE004, Mittweida
- Serbia (5):
  - RS002, Belgrade
  - RS003, Belgrade
  - RS004, Belgrade
  - RS005, Belgrade
  - RS001, Kragujevac
- Slovakia (4):
  - SK004, Bratislava
  - SK001, Domaša
  - SK003, Levice
  - SK002, Rimavská Sobota

REFERENCES:
- [Derived] Christensen MC, Sluth LB, McIntyre RS. Validation of the University of California San Diego Performance-based Skills Assessment (UPSA) in major depressive disorder: Replication and extension of initial findings. J Affect Disord. 2019 Feb 15;245:508-516. doi: 10.1016/j.jad.2018.11.034. Epub 2018 Nov 5. PMID 30439678
- See also: EMA EudraCT Results: 2014-000230-34 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-000230-34/results